CLINICAL TRIAL: NCT04303858
Title: An Open-Label, Multicenter, Randomized, Dose-Escalation and Extension, Phase IA/IB Study to Evaluate Safety and Anti-Tumor Activity of RO7284755, A PD-1 Targeted IL-2 Variant (IL-2V) Immunocytokine, Alone or in Combination With Atezolizumab in Participants With Advanced and/or Metastatic Solid Tumors
Brief Title: A Study to Evaluate Safety and Anti-Tumor Activity of Eciskafusp Alfa (RO7284755) Alone or in Combination With Atezolizumab in Participants With Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP41628; 2019-004022-25 (EudraCT Number); 2023-503749-76-00 (EU CTIS Number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eciskafusp Alfa as a Single Agent (Experimental): Part 1: Dose-escalation of eciskafusp alfa as a single agent. eciskafusp alfa will be either an intravenous administration (IV) or subcutaneous administration (SC) in multiple-ascending doses.
  Interventions: Drug: Eciskafusp Alfa
- Eciskafusp Alfa in Combination with Atezolizumab (Experimental): Part 2: Dose-escalation of eciskafusp alfa in combination with atezolizumab.
  Interventions: Drug: Eciskafusp Alfa; Drug: Atezolizumab
- Eciskafusp Alfa as a Single Agent and/or with Atezolizumab (Experimental): Part 3: Extension of eciskafusp alfa as a single agent and/or in combination with atezolizumab.
  Interventions: Drug: Eciskafusp Alfa; Drug: Atezolizumab

INTERVENTIONS:
Drug: Eciskafusp Alfa — Participants will be administered eciskafusp alfa in different schedules.
  Other Names: RO7284755
Drug: Atezolizumab — Participants will be administered 1200 mg of atezolizumab once every 3 weeks.
  Other Names: Tecentriq
  Arms: Eciskafusp Alfa as a Single Agent and/or with Atezolizumab; Eciskafusp Alfa in Combination with Atezolizumab

SUMMARY:
This is an entry-into-human study and will assess the effects of eciskafusp alfa (RO7284755) as a single agent and in combination with atezolizumab in adult participants with solid tumors considered responsive to checkpoint inhibition blockade. The maximum duration in the study for each participant will be up to 28 months.

DETAILED DESCRIPTION:
The study consists of three parts: dose-escalation of eciskafusp alfa as a single agent (Part 1), dose-escalation of eciskafusp alfa in combination with atezolizumab (Part 2), and extension of eciskafusp alfa as a single agent and/or in combination with atezolizumab (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced/unresectable or metastatic disease
* No standard of care (SoC) (approved) treatments are available for the participant, or the participant cannot tolerate such treatments
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group Performance Status 0 to 1
* Life expectancy of >=12 weeks
* Consent to provide an archival tumor tissue sample
* Adequate cardiovascular, hematological, coagulative, hepatic and renal function

Exclusion Criteria:

* Rapid disease progression or suspected hyperprogression or threat to vital organs or critical anatomical sites requiring urgent alternative medical intervention
* Untreated central nervous system (CNS) metastases
* Treated asymptomatic CNS metastases
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >= 2 weeks before Cycle1 Day 1 (C1D1)
* Active or history of carcinomatous meningitis/leptomeningeal disease
* Uncontrolled tumor-related pain or symptomatic hypercalcemia
* Concurrent second malignancy
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
* Episode of significant cardiovascular/cerebrovascular acute disease within 28 days before study treatment administration
* Active or uncontrolled infections
* Known HIV infection
* Hepatitis B virus (HBV) or hepatitis C virus infection
* Adverse events related to any prior radiotherapy, chemotherapy, targeted therapy, CPI therapy or surgical procedure must have resolved to Grade <=1, except alopecia Grade 2 peripheral neuropathy, and hypothyroidism and/or hypopituitarism on a stable dosage of hormone replacement therapy
* Participants with bilateral pleural effusion
* Major surgery or significant traumatic injury < 28 days before study treatment administration or anticipation of the need for major surgery during study treatment
* Known allergy or hypersensitivity to any component of the formulations of the IMPs to be administered, including but not limited to hypersensitivity to Chinese hamster ovary cell products or other recombinant or humanized antibodies
* History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins
* Previous treatment with Interleukin-2 (IL-2)/Interleukin-5 (IL-15)-like cytokines. IL-2/IL-15 use as an adjunct treatment component for adoptive cell therapy is permitted. In Part 3, patients who have received adoptive cell therapy such as tumor-infiltrating lymphocytes (TIL) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events in Part 1 and Part 2 | From randomization until end of Part 1 and Part 2 (up to approximately 1.5 months)
  An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. All AE events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Percentage of Participants with Dose-Limiting Toxicities in Part 1 and Part 2 | From randomization up to day 14 (Part 1) or day 28 (Part 2)
  A DLT is defined as a clinically significant AE (classified according to the NCI CTCAE version 5) or significant laboratory abnormality that occur during the DLT assessment periods, during Part 1 and Part 2 only, and is considered by the Investigator to be related to eciskafusp alfa or to the combination of eciskafusp alfa and atezolizumab. In Part 2, expected toxicities that are, in the opinion of the Investigator, entirely attributable to atezolizumab, will not be considered DLTs.
Investigator Assessed Objective Response Rate according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Part 3 | From start of extension phase until disease progression, drug discontinuation, withdrawal or death (up to approximately 26 months)
  Objective response rate (ORR) was defined as the percentage of participants with investigator-assessed objective response of complete response (CR) or partial response (PR). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions).
Recommended Dose for Extension (RDE) of Eciskafusp Alfa in Parts 1 and 2 | From randomization up to day 14 (Part 1) or day 28 (Part 2)

SECONDARY OUTCOMES:
Investigator Assessed Objective Response Rate according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Parts 1 and 2 | From randomization until end of Part 1 and Part 2 (up to approximately 1.5 months)
  ORR was defined as the percentage of participants with investigator-assessed objective response of complete response (CR) or partial response (PR). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions).
Percentage of Participants with Adverse Events in Part 3 | From start of extension phase until disease progression, drug discontinuation, withdrawal or death (up to approximately 26 months)
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. All AE events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Disease Control Rate in Part 3 | From start of extension phase until disease progression, drug discontinuation, withdrawal or death (up to approximately 26 months)
  The disease control rate was defined as proportion of participants being either responder or in 'stable disease' (SD). To classify a response as SD, measurements will have to be classified as stable (according to RECIST v1.1) at least once at a minimum of 4 weeks after study entry.
Duration of Response in Part 3 | From start of extension phase until disease progression, drug discontinuation, withdrawal or death (up to approximately 26 months)
  Duration of response will be calculated for 'responder' participants (i.e. best [confirmed] overall response of CR or PR) and will be defined as the time from first occurrence of a documented response until the time of documented disease progression or death (death within 30 days from last study treatment) from any cause, whichever occurs first.
Progression-free survival (PFS) in Part 3 | From start of extension phase until disease progression, drug discontinuation, withdrawal or death (up to approximately 26 months)
  Progression-free survival was defined as the time from first dose of study treatment to the first occurrence of documented disease progression (based on RECIST 1.1 Investigator's assessment) or death from any cause, whichever occurs first.
Change from Baseline in Antidrug Antibody (ADA) to Eciskafusp Alfa | Up to 28 months
Percentage of Partcipants with ADAs to Eciskafusp Alfa | Up to 28 months
Area Under the Curve (AUC) for Eciskafusp Alfa | Predose, C1 Days 1, 2, 3, 5, 8, 9, 10, 12, 15, 16, 17, and 19; C2 Days 1, 2, 8, 9, 10, 12, 15, and 16; C3 Days 1, 2, 3, and 8; C4 Days 1 and 2; C5 Days1, 2, and 8; and days 1 and 2 for any subsequent cycles (Up to 28 months)
Minimum Concentration (Cmin) for Eciskafusp Alfa | Predose, C1 Days 1, 2, 3, 5, 8, 9, 10, 12, 15, 16, 17, and 19; C2 Days 1, 2, 8, 9, 10, 12, 15, and 16; C3 Days 1, 2, 3, and 8; C4 Days 1 and 2; C5 Days1, 2, and 8; and days 1 and 2 for any subsequent cycles (Up to 28 months)
Maximum Concentration (Cmax) for Eciskafusp Alfa | Predose, C1 Days 1, 2, 3, 5, 8, 9, 10, 12, 15, 16, 17, and 19; C2 Days 1, 2, 8, 9, 10, 12, 15, and 16; C3 Days 1, 2, 3, and 8; C4 Days 1 and 2; C5 Days1, 2, and 8; and days 1 and 2 for any subsequent cycles (Up to 28 months)
Clearance (CL) for Eciskafusp Alfa | Predose, C1 Days 1, 2, 3, 5, 8, 9, 10, 12, 15, 16, 17, and 19; C2 Days 1, 2, 8, 9, 10, 12, 15, and 16; C3 Days 1, 2, 3, and 8; C4 Days 1 and 2; C5 Days1, 2, and 8; and days 1 and 2 for any subsequent cycles (Up to 28 months)
Volume of Distribution at Steady-State Conditions (Vss) for Eciskafusp Alfa | Predose, C1 Days 1, 2, 3, 5, 8, 9, 10, 12, 15, 16, 17, and 19; C2 Days 1, 2, 8, 9, 10, 12, 15, and 16; C3 Days 1, 2, 3, and 8; C4 Days 1 and 2; C5 Days1, 2, and 8; and days 1 and 2 for any subsequent cycles (Up to 28 months)
Percentage of Immune and Tumor Cells with Positive Programmed Cell Death-1 (PD-1) and Programmed Cell Death-Ligand 1 (PD-L1) Expression in the Tumor Microenvironment (TME) | Baseline
Percentage of Immune Cells with CD8+ PD1+ and CD8+ PD1+ TCF7+ Expression | Baseline
Blood Tumor Mutational Burden | Baseline
  Blood tumor mutational burden is defined as the number of genetic mutations per megabase (1,000,000 bases).
Change from Baseline in Percentage of Immune Cell Subsets | Baseline to End of Treatment (up to approximately 28 months)
  Immune cells include NK, CD8, and Treg cells
Change from Baseline in Percentage of Immune Markers | Baseline to End of Treatment (up to approximately 28 months)
  Immune markers include PD-1, PD-L1, sCD25, cytokines, etc...

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Denmark (2):
  - Herlev Hospital, Herlev
  - Rigshospitalet, København Ø
- Netherlands (2):
  - NKI/AvL, Amsterdam
  - Erasmus MC, Rotterdam
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Warsaw
- Spain (4):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No